CLINICAL TRIAL: NCT02127255
Title: Acupuncture for Chemical Therapy Induced Nausea and Vomiting: a Cross-over Trail
Acronym: ACTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yutong Fei, Associate research fellow, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EBM@BUCM-1; Z111107054511086 (Other Grant/Funding Number: Beijing Nova Program)
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: chemotherapy; nausea; vomiting; cancer
MeSH Terms: conditions — Vomiting; Nausea; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Acupuncturist 1) (Active Comparator): Manual acupuncture implemented by acupuncturist 1 (clinical experience >15 years)
  Interventions: Procedure: Manual acupuncture implemented by acupuncturist 1
- B (Acupuncturist 2) (Active Comparator): Manual acupuncture implemented by acupuncturist 2 (clinical experience < 5 years)
  Interventions: Procedure: Manual acupuncture implemented by acupuncturist 2

INTERVENTIONS:
Procedure: Manual acupuncture implemented by acupuncturist 1 — Manual acupuncture once per day. Acupuncture treatment regimens (acupoints, needling methods, needle retention time) were decided by acupuncturist 1 according to the syndrome differentiation of patients. Acupuncturist 1 has to have more than 15 years of acupuncture clinical practice experience.
  Other Names: Traditional manual acupuncture; Traditional acupuncture
  Arms: A (Acupuncturist 1)
Procedure: Manual acupuncture implemented by acupuncturist 2 — Manual acupuncture given by acupuncturist 2 once per day. Acupuncture treatment regimens (acupoints, needling methods, needle retention time) were decided by acupuncturist 1 according to the syndrome differentiation of patients. Acupuncturist 2 has to have less than 5 years of acupuncture clinical practice experience.
  Other Names: Traditional manual acupuncture; Traditional acupuncture
  Arms: B (Acupuncturist 2)

SUMMARY:
This is a randomized, controlled cross-over trial. The hypothesis of this study is that the differences in manual acupuncture manipulation can impact clinical effect though the acupuncturists follow the same needling regimen. In this study, acupuncturist 1 (clinical experience >15 years) and acupuncturist 2 (<5 years) will give treatments to cancer patients receiving cisplatin chemotherapy (n=36) for at least two continuous cycles, once per day, 5 days per cycle. Acupuncturist 1 determines all the treatment regimens (selection of acupoints and methods of needling manipulation, needle retention time). Randomly, half of the patients will receive treatments from acupuncturist 1 in the first treatment cycle and from acupuncturist 2 in the second cycle; while the other half will be treated in other way round. There is a washout period (21 days) between two cycles. The needling manipulation of two acupuncturists will be measured objectively during treatments. The clinical effect will be measured by the control of vomiting and nausea during and after chemotherapy treatments.

DETAILED DESCRIPTION:
This is a randomized, controlled cross-over trial. The hypothesis of this study is that the differences in manual acupuncture manipulation can impact clinical effect though the acupuncturists follow the same needling regimen. In this study, acupuncturist 1 (clinical experience >15 years) and acupuncturist 2 (<5 years) will give treatments to cancer patients receiving cisplatin chemotherapy (n=36) for at least two continuous cycles, once per day, 5 days per cycle. Acupuncturist 1 determines all the treatment regimens (selection of acupoints and methods of needling manipulation, needle retention time). Randomly, half of the patients will receive treatments from acupuncturist 1 in the first treatment cycle and from acupuncturist 2 in the second cycle; while the other half will be treated in other way round. There is a washout period (21 days) between two cycles. The needling manipulation of two acupuncturists will be measured objectively during treatments. The clinical effect will be measured by the control of vomiting and nausea during and after chemotherapy treatments. The manual manipulation of two acupuncturists will be recorded by device Acusensor.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cancer
* Must receive cancer chemotherapy containing cisplatin
* Able to complete at least two continuous chemotherapy treatment cycles
* Karnofsky performance status grade ≥60
* Must use 5-TH receptor antagonists as an antiemetic drug in the chemotherapy duration

Exclusion Criteria:

* Concurrent neoplasms or illness that induces nausea independent of chemotherapy
* Receiving radiotherapy
* Received acupuncture treatments for other conditions less than 4 weeks before chemotherapy treatment
* Severe infection
* Severe heart, liver, kidney and brain diseases
* Unconsciousness
* Psychosis
* Language barriers
* Cardiac pacemaker
* Radiotherapy or hormone therapy during chemotherapy treatments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
NCI nausea and vomiting rating scale | day1-8 on each study period

SECONDARY OUTCOMES:
Rhodes Scale | day1-5 on each study period
global assessment on effectiveness by patients (VAS) | day 5 on each study period
patients' confidence towards acupuncture treatment(VAS) | day 1,5 on each study period
global satisfaction for acupuncture treatments | day 5 on each study period
Acupuncture Expectancy Scale (AES) | day 1, 3, 5 on each study period

OTHER OUTCOMES:
patient communication satisfaction scale | day 5 on each study period
Acupuncture related adverse events | day 1-5 each study period
  faintng during acupuncture treatment, sticking of needle, bleeding in the needling hole, broken needles
Adverse events (not acupuncture treatment specified) | day 1-5 each study period
Needling manipulation parameters | day 1-5 each study period
  Displacement Frequency (Hz) Displacement Amplitude (pk-pk) Rotation Frequency (Hz) Rotation Amplitude (pk-pk)

CONTACTS AND LOCATIONS:
Overall Officials: Yutong Fei, MD, Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided